CLINICAL TRIAL: NCT05819944
Title: A Trial Evaluating Novel Technologies for the Diagnosis of Asthma
Brief Title: A Trial Evaluating Novel Technologies for the Diagnosis of Asthma The LUNG-TECH Trial
Acronym: LUNG-Tech
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHU/2022/36
Record Dates: First submitted 2023-02-20; First posted 2023-04-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Pathway 1- Diagnostic case control study undertaken in a secondary care population: evaluates whether the technology can distinguish between people with asthma and healthy volunteers, and other respiratory conditions in a well characterised secondary care population;
- Pathway 2- Prospective diagnostic study undertaken in a primary care population: assesses whether the technology can accurately diagnose asthma (either independently or alongside current diagnostic tests) in a primary care population of patients where there is a clinical suspicion of asthma;
- Pathway 3- A phenotypic characterisation study undertaken in participants with confirmed asthma: explores the ability of the technology to identify clinically important phenotypic characteristics which are difficult to measure in primary care and/or significantly impact on patient management and treatment;

SUMMARY:
This trial aims to evaluate novel diagnostic technologies for asthma in 3 different pathways providing the necessary evidence-base to allow adoption into clinical practice:

* Pathway 1 evaluates whether the technology can distinguish between people with asthma and healthy volunteers, and other respiratory conditions in a well characterised secondary-care population and whether the parameters they measure correlate with the current standard diagnostic tests;
* Pathway 2 assesses whether the technology can accurately diagnose asthma (either independently or alongside current diagnostic tests) in a primary care population of patients where there is a clinical suspicion of asthma;
* Pathway 3 explores the ability of the technology to identify clinically important phenotypic characteristics which are difficult to measure in primary care and/or significantly impact on patient management and treatment

The novel technology and devices will be entered into the pathway most suited to their stage of development, with this study design also allowing information collected for participants with a confirmed diagnosis of asthma in pathways 1 or 2 to be included in pathway 3. Participants will undergo the investigations currently used to diagnose asthma as well as using the novel devices being investigated in the relevant pathway.

DETAILED DESCRIPTION:
This trial aims to evaluate novel diagnostic technologies for asthma in 3 different pathways providing the necessary evidence-base to allow adoption into clinical practice.

Pathway 1: Diagnostic case control study undertaken in a secondary care population

This will assess whether the novel technology can differentiate asthma from other respiratory conditions and from healthy volunteers, and whether the parameters they measure correlate with the current standard diagnostic tests (in line with the NICE algorithm) including those methods assessing airway inflammation and disease severity. Assessment of safety and acceptability of the technology will also be undertaken. We will invite patients who have asthma, other respiratory conditions and people who do not have any breathing problems to take part. It will be a single visit and all eligible participants will perform informed consent, and will then have baseline characteristics recorded, along with past medical history and demographical information. Participants will undergo the investigations currently used for the asthma diagnostic work-up in routine care. This will include spirometry, airway inflammation measurements (using FeNO), oscillometry and blood tests (where these have not been taken in the preceding 12 months). Participants will also be asked to use the novel device(s) currently being tested in this pathway. All participants will be asked to answer a questionnaire about how easy they found each test to use.

Pathway 2: Prospective diagnostic study undertaken in a primary care population

This study will assess whether the novel technology can be used to accurately diagnose asthma independently or whether it can be used alongside current diagnostic tests to improve the diagnostic pathway for patients with asthma. Acceptability of the novel device to patients and HCPs will be measured and the feasibility of using the novel device in the clinical pathway will be assessed. Participants with a clinical suspicion of asthma presenting with ≥1 symptom suggestive of asthma identified will be identified either from GP practices or patients presenting to the Portsmouth asthma service with diagnostic uncertainty.

Participants will undergo a comprehensive specialist assessment in line with the NICE asthma diagnostic algorithm mirroring our routine standard of care. This phase will consist of 3-4 visits depending on the results.

* Visit 0- informed consent will be taken and an initial clinical assessment will be undertaken including- demographics, symptom/asthma and other medical history review, medication review and co-morbidity assessment. Participants will complete a series of questionnaires assessing disease control, quality of life and co-morbidities. They will be provided with a peak flow meter and asked to keep a diary for 2-weeks.
* Visit 1- all participant's will undergo a comprehensive work-up including spirometry and oscillometry (pre and post bronchodilator), FeNO, blood tests and skin prick testing. They will also be asked to use the novel device and complete a short visual analogue scale questionnaire to explore the ease of use and acceptability of the device as a diagnostic test. Where a diagnosis of asthma can be made based on the testing done, participants will be commenced on treatment with an inhaled corticosteroid treatment (in line with our regional guidelines) and will be followed-up in 4-weeks from starting treatment. Where a diagnosis cannot be made, participants will be invited back to undergo a Methacholine challenge test.
* Visit 2 (only required for participants undergoing a Methacholine challenge test)- a diagnosis of asthma will either be confirmed, excluded or a treatment trial will be required. Where asthma is confirmed or a trial of treatment recommended, participants ill be commenced on treatment with an inhaled corticosteroid treatment (in line with our regional guidelines) and will be followed-up in 4-weeks from starting treatment.
* Visit 3: Further clinical assessment to assess response to treatment. Where needed diagnosis will be confirmed or excluded. Where asthma is confirmed all participants will be provided with an asthma self-management plan (if this has not happened in an earlier visit).

All participants will have asthma either confirmed or excluded by the end of their study visits with treatment commenced where appropriate. A report will be issued to both themselves and their GP outlining the results of their investigations and any ongoing management recommendations.

Pathway 3: A phenotypic characterisation study undertaken in participants with confirmed asthma

This study will assess the ability of the novel device to identify clinically important phenotypic characteristics which are difficult to measure in primary care and/or significantly impact on patient management and treatment. Important phenotypic characteristics include: T2 inflammation; Small airways dysfunction; Overlapping Breathing Pattern Disorder.

Participants with confirmed asthma (including those identified from Pathways 1 and 2) will be recruited and undergo an enhanced characterisation, including detailed lung function testing, biomarker assessment for T2 airway inflammation and co-morbidity questionnaires. This phase can run in parallel to Pathways 1 and 2 if necessary and where these investigations have already been undertaken in earlier phases, they will not be repeated with the earlier results being used.

All participants and healthcare professionals involved in the study will also be asked to complete a short visual analogue scale questionnaire to explore the ease of use and acceptability of the device as a diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis confirmed by a specialist supported by any of the following within the last 5-years: i) Evidence of variable and/or reversible airflow obstruction
* FEV1/FVC ratio <70% on spirometry with FEV1 ≥12% and 200 ml increase post-BD or
* FEV1 variability ≥20% between clinic visits within 12-months or
* R5-R20 ≥0.1kPa/(L/s) with ≥40% improvement post-BD or ii) Evidence of significant peak expiratory flow (PEF) variability
* ≥ 20% PEF variability iii) Evidence of airway hyperresponsiveness (AHR)
* Positive methacholine challenge test (PD20 ≤8mg/ml) or equivalent iv) Evidence of T2 airway inflammation
* FeNO ≥40ppb

  * Poor disease control evidenced by an ACQ-6 score ≥1.5
  * Not on a biologic therapy for severe asthma

Exclusion Criteria:

* • Known clinically significant chest wall, neuromuscular, cardiac or other co-morbidity or abnormality that would affect spirometry and/or other measures of lung function/inflammation (in the opinion of the investigator)

  * Respiratory tract infection/exacerbation of respiratory condition requiring systemic corticosteroids and/or antibiotic treatment within the last 2 weeks
  * Current smokers or Ex-smokers with >20 PYH (other than COPD and asthma with significant smoking history group)
  * The participant is unable to provide informed consent or is unable to complete the study procedures

Healthy Volunteers:

* No current clinical diagnosis of (or treatment for) a respiratory disease and no treatment for a respiratory tract Infection within the last 6 months
* Never smoker or ex-smoker with ≤10 pack-years smoking history, and stopped smoking at least 6-months prior to enrolment
* Non-obstructive spirometry

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from outpatient and community respiratory clinics and local GP practices, with study activity taking place in both primary and secondary care.
Sampling Method: Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pathway 1 | 3 months
  The difference in each of the parameters (and combinations of these parameters), measured using the novel technology in patients with asthma, other respiratory conditions (COPD, BPD, bronchiectasis), and healthy volunteers
  As this is a pathway trial, it is not possible to define all of the parameters proactively as the novel devices included with the pathway will increase/change. This would be updated via amendments which will include devices and parameters
Pathway 2 | 6 months
  Compare each device-specific parameter measured using the novel technology (and combinations of these parameters) between asthma, other respiratory conditions (COPD, BPD, bronchiectasis), and healthy volunteers
  Compare levels of device-specific parameters independently or in combination, that optimally discriminate between asthma, other respiratory conditions (COPD, BPD, bronchiectasis), and healthy volunteers.
  As this is a pathway trial, it is not possible to define all of the parameters proactively as the novel devices included with the pathway will increase/change. This would be updated via amendments which will include devices and parameters
Pathway 3 | 6 months
  To assess the associations between each of the parameters (and combinations of these parameters) measured by the novel technology and the presence of:
  * T2 inflammation (defined by FeNO ≥40ppb and/or blood eosinophils ≥0.3x109/L)
  * SAD (IOS R5-R20 ≥0.1kPa/(L/s) and/or HRCT chest evidence of gas trapping
  * BPD defined by a BPAT score ≥4 or a specialist diagnosis
  As this is a pathway trial, it is not possible to define all of the parameters proactively as the novel devices included with the pathway will increase/change. This would be updated via amendments which will include devices and parameters

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dr Brown, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No